CLINICAL TRIAL: NCT07338071
Title: Antithrombotic Therapy at the End of Life: The PEACE Study
Acronym: PEACE
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Ospedale Cristo Re - Roma (Unknown); San Giovanni Addolorata Hospital (Other)
Responsible Party: Principal Investigator, Pola Roberto, Prof., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: ID 3722
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Palliative Care
Keywords: antithrombotic therapy; end of life; palliative care
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: antithrombotic drugs — use of antithrombotic drug

SUMMARY:
"Antithrombotic Therapy at the End of Life: The PEACE Study" is a multicenter, non-profit, cross-sectional observational study. In the absence of shared guidelines, therapeutic decisions on antithrombotic drugs vary significantly according to healthcare professional training and national context, resulting in marked variability in prescribing practices. This study aims to describe the prevalence of antithrombotic prescriptions in patients referred to Palliative Care.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) hospitalized and referred to Palliative Care (home-based or residential) at the discretion of the attending physician.
* Signed informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sample will consist of hospitalized patients referred to a Palliative Care pathway
Sampling Method: Non-Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence of antithrombotic drug use | at enrollment
  Calculation of the prevalence of antithrombotic drug use in hospitalized patients referred to Palliative Care pathway.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No